CLINICAL TRIAL: NCT06018870
Title: MRI Contrast Clearance Analysis for Prediction of Grading and Genotyping in Gliomas
Brief Title: MRI Contrast Clearance Analysis for Glioma Grading and Genotyping
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Daping Hospital and the Research Institute of Surgery of the Third Military Medical University (Other)
Responsible Party: Principal Investigator, Weiguo Zhang, Chief of radiology department, Daping Hospital and the Research Institute of Surgery of the Third Military Medical University
Other Study IDs: 2023183
Record Dates: First submitted 2023-08-24; First posted 2023-08-31 (Actual); Last update posted 2023-08-31 (Actual); Status verified 2023-08

CONDITIONS: Glioma
Keywords: Glioma
MeSH Terms: conditions — Glioma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Gliomas are the most common primary brain tumor. Gliomas with different grades have different clinical behaviors that determine treatment planning and patient prognosis in clinical practice. In the 2021 World Health Organization (WHO) classification of tumors for the central nervous system, glioma genotyping was considered the most relevant information for neuroradiologists. The isocitrate dehydrogenase (IDH) genotype and 1p/19q codeletion status are two essential molecular markers that divide glioma into three groups: IDH wild-type, IDH mutant with 1p/19q non-codeletion, and IDH mutant with 1p/19q codeletion.

MRI contrast clearance analysis (CCA) is based on T1 delayed-contrast subtraction map, Blue/tumor regions in CCA represent efficient clearance of contrast from the tissue (delayed signal<early signal), while red/nontumor regions in CCA represent contrast accumulation (delayed signal>early signal).

However, there are not any reports on the role of MRI CCA in glioma grading and genotyping, Thus, We hypothesized that the proportion of blue/red region and their histogram analyses, which could be acquired for predicting IDH genotypes and 1p/19q codeletion in gliomas, and to assess the application of CCA in glioma grading.

DETAILED DESCRIPTION:
This is a single-center bidirectional cohort study. The subjects of this study were patients diagnosed as glioma by pathological biopsy. Patients with suspicious mass will be performed extra 30 and 60 min after contrast agent application delayed T1-weighted sequences as same as before. Then enter the next experimental stage. (1) Image format conversion; (2) Registration;(3) Subtraction;(4) ROI segmentation;(5) ROI histogram analyses. Histogram parameters of blue and red ROI includes 1st、10th 、90th and 99th percentiles, mean, median, variance, skewness, and kurtosis.

Finally, statistical methods were used to determine whether those parameters was statistically significant for IDH mutation status、1p/19q codeletion status and tumor grading.

ELIGIBILITY:
Inclusion Criteria:

* Patients with brain space -occupying lesions, have not yet undergone antitumor therapy;
* MRI with T1-contract delayed sequence was performed less than 2 weeks before surgery;
* Definite histopathologic diagnosis of glioma.

Exclusion Criteria:

* WHO 1 gliomas and other non-glioma brain tumors;
* Poor image quality and heavy artifact affect the subsequent image processing.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The subjects are not restricted by gender and age. For details, please refer to the "criteria" column.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of bule/red ROI | Through study completion, an average of 1 year
  The common vessels morphology in the blue region was undamaged vessel lumens which exists in active tumor, while vessels in the red regions presented different stages of vessel necrosis.
Histogram of bule/red ROI | Through study completion, an average of 1 year
  The bule and red ROI from CCA histogram analysis included1st、10th 、90th and 99th percentiles, mean, median, variance, skewness, and kurtosis.

CONTACTS AND LOCATIONS:
Locations (1):
- Sang Zifan, Chongqing, Chongqing Municipality, China